CLINICAL TRIAL: NCT04606654
Title: Effects of Handgrip Training With and Without Blood Flow Restriction in Relation to Gender Among Healthy Young Adults
Brief Title: Handgrip Training With and Without Blood Flow Restriction in Relation to Gender Among Healthy Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/788 Arva Naeem
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Sports Physical Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Handgrip strength training with Blood flow restriction (Experimental): Three sessions per week will be given to individual subject. and training will be with Blood flow restriction.
  Subjects will be followed for two weeks for;
  * Hand grip strength
  * Forearm circumference
  Interventions: Other: Handgrip strength training with Blood flow restriction
- Handgrip strength training without Blood flow restriction (Active Comparator): Three sessions per week will be given to individual subject and training will be without Blood flow restriction.
  Subjects will be followed for two weeks for;
  * Hand grip strength
  * Forearm circumference
  Interventions: Other: Handgrip strength training without Blood flow restriction

INTERVENTIONS:
Other: Handgrip strength training without Blood flow restriction — Participants of this group will get exercise training through hand grip strengthener and DMOOSE fitness resistance bar. Participants will contract his/her forearm at a rate of 15 times/min (1 contraction every 4 sec). The subjects will train for 20 min, 3 days per week for 2 weeks (total 6 sessions), under the supervision of a principle investigator. Participants will be allowed to take 1 min rest periods, after the completion of 5 minutes of training.
  Arms: Handgrip strength training without Blood flow restriction
Other: Handgrip strength training with Blood flow restriction — Participants of this group will get exercise training through hand grip strengthener and DMOOSE fitness resistance bar. Participants will contracts his/her forearm at a rate of 15 times/min (1 contraction every 4 sec). The subjects will train for 20 min, 3 days per week for 2 weeks (total 6 sessions), under the supervision of a principle investigator. Participants will be allowed to take 1 min rest periods, after the completion of 5 minutes of training. However, for one of the limbs the pneumatic blood pressure cuff will be placed on the upper arm, 4 cm proximal to the ante-cubital fossa. The decision which arm would receive the occlusion during training will be randomized to avoid a dominant or non-dominant hand bias. During experimental group training blood pressure cuff will be partially inflated (80 mmHg) to ensure venous occlusion. Participants will be allowed to take 1 min rest periods, after the completion of 5 minutes of training while the cuff remained inflated.
  Arms: Handgrip strength training with Blood flow restriction

SUMMARY:
In this study Investigator will determine the effects of blood flow restriction training on hand grip strength using hand held dynamometer among healthy young adults and investigator also see effects of blood flow restriction training on forearm circumference using weighted measuring tape among healthy young adults along with correlation of male and female population following blood flow restriction training among healthy young adults.

DETAILED DESCRIPTION:
(A randomized control trial will be conducted in Foundation University Institute of Rehabilitation Sciences on 56 healthy young adults. Study will be conducted in 6 months (May 2020 to December 2020). Healthy young adults of both genders between 20-40 years of age will be included in the study. Adults with any diagnosed cardiovascular, metabolic, orthopedic or neurological disease, active/ongoing infection, recent history of upper extremity fracture or history of vascular medication will not be included in this study. The outcome variables will be hand grip strength measured through hydraulic hand held dynamometer and forearm circumference through anthropometric measuring tape.After assessment and screening, subjects will be randomly allocated in Control group "A" receiving low intensity strength training and Interventional group "B" receiving blood flow restriction training along with low intensity strength training via lottery method.Each participant will receive three sessions per week for two consecutive weeks making 6 treatment sessions in total. The outcome variables will be assessed at the start of 1st session and then at 6th session. To carry out the anthropometric assessment, anthropometric tape for circumference measurements, a digital scale for measuring weight and a stadiometer to measure height will be used.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults of sedentary lifestyle
* Young healthy adults following 6 minutes' Walk test
* Young healthy adults following YMCA 3 minutes Step test

Exclusion Criteria:

* Any diagnosed cardiovascular, metabolic, orthopaedic or neurological disease
* Active/ongoing infection
* Recent history of upper extremity fracture
* History of vascular medication

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Hand grip strength | 8 weeks
  Changes from the baseline, To measure hand grip strength through Hydraulic Hand held Dynamo-meter. It will be measured in pounds
Forearm circumference | 8 weeks
  After strength training forearm circumference through anthropometric measuring tape will be measured in inches by inches measuring tape.

CONTACTS AND LOCATIONS:
Overall Officials: Suhail Karim, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Foundation University Institute of Rehabilitation Sciences, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hughes L, Paton B, Rosenblatt B, Gissane C, Patterson SD. Blood flow restriction training in clinical musculoskeletal rehabilitation: a systematic review and meta-analysis. Br J Sports Med. 2017 Jul;51(13):1003-1011. doi: 10.1136/bjsports-2016-097071. Epub 2017 Mar 4. PMID 28259850
- [Background] Lixandrao ME, Ugrinowitsch C, Berton R, Vechin FC, Conceicao MS, Damas F, Libardi CA, Roschel H. Magnitude of Muscle Strength and Mass Adaptations Between High-Load Resistance Training Versus Low-Load Resistance Training Associated with Blood-Flow Restriction: A Systematic Review and Meta-Analysis. Sports Med. 2018 Feb;48(2):361-378. doi: 10.1007/s40279-017-0795-y. PMID 29043659
- [Background] Cristina-Oliveira M, Meireles K, Spranger MD, O'Leary DS, Roschel H, Pecanha T. Clinical safety of blood flow-restricted training? A comprehensive review of altered muscle metaboreflex in cardiovascular disease during ischemic exercise. Am J Physiol Heart Circ Physiol. 2020 Jan 1;318(1):H90-H109. doi: 10.1152/ajpheart.00468.2019. Epub 2019 Nov 8. PMID 31702969
- [Background] Pearson SJ, Hussain SR. A review on the mechanisms of blood-flow restriction resistance training-induced muscle hypertrophy. Sports Med. 2015 Feb;45(2):187-200. doi: 10.1007/s40279-014-0264-9. PMID 25249278
- [Background] Sato, Y., The history and future of KAATSU training. International Journal of KAATSU Training Research, 2005. 1(1): p. 1-5.
- [Background] Yasuda, T., et al., Use and safety of KAATSU training: Results of a national survey in 2016. International Journal of KAATSU Training Research, 2017. 13(1): p. 1-9.
- [Background] O'Brien, L. Blood Flow Restriction Therapy. 2020 [cited 2020; Available from: https://members.physio-pedia.com/learn/blood-flow-restriction-therapy/.
- [Background] Cardoso RK, Araujo AM, Del Vechio FB, Bohlke M, Barcellos FC, Oses JP, de Freitas MP, Rombaldi AJ. Intradialytic exercise with blood flow restriction is more effective than conventional exercise in improving walking endurance in hemodialysis patients: a randomized controlled trial. Clin Rehabil. 2020 Jan;34(1):91-98. doi: 10.1177/0269215519880235. Epub 2019 Oct 11. PMID 31603002
- [Background] Jessee MB, Dankel SJ, Buckner SL, Mouser JG, Mattocks KT, Loenneke JP. The Cardiovascular and Perceptual Response to Very Low Load Blood Flow Restricted Exercise. Int J Sports Med. 2017 Jul;38(8):597-603. doi: 10.1055/s-0043-109555. Epub 2017 Jun 26. PMID 28651256
- [Background] Brandner CR, Kidgell DJ, Warmington SA. Unilateral bicep curl hemodynamics: Low-pressure continuous vs high-pressure intermittent blood flow restriction. Scand J Med Sci Sports. 2015 Dec;25(6):770-7. doi: 10.1111/sms.12297. Epub 2014 Jul 23. PMID 25055880
- [Background] Araujo JP, Silva ED, Silva JC, Souza TS, Lima EO, Guerra I, Sousa MS. The acute effect of resistance exercise with blood flow restriction with hemodynamic variables on hypertensive subjects. J Hum Kinet. 2014 Nov 12;43:79-85. doi: 10.2478/hukin-2014-0092. eCollection 2014 Sep 29. PMID 25713647
- [Background] Centner C, Wiegel P, Gollhofer A, Konig D. Correction to: Effects of Blood Flow Restriction Training on Muscular Strength and Hypertrophy in Older Individuals: A Systematic Review and Meta-Analysis. Sports Med. 2019 Jan;49(1):109-111. doi: 10.1007/s40279-018-1013-2. PMID 30414044
- [Background] Jacobson, J., et al., Blood Flow Restriction Training in Clinical Musculoskeletal Rehabilitation: A Critically Appraised Paper. International Journal of Athletic Therapy and Training, 2020. 1(aop): p. 1-4.
- [Background] Pope ZK, Willardson JM, Schoenfeld BJ. Exercise and blood flow restriction. J Strength Cond Res. 2013 Oct;27(10):2914-26. doi: 10.1519/JSC.0b013e3182874721. PMID 23364292
- [Background] Credeur DP, Hollis BC, Welsch MA. Effects of handgrip training with venous restriction on brachial artery vasodilation. Med Sci Sports Exerc. 2010 Jul;42(7):1296-302. doi: 10.1249/MSS.0b013e3181ca7b06. PMID 20019641
- [Background] https://www.sralab.org/. 6 Minute Walk Test. 2020 2020 [cited 2020; Available from: https://www.sralab.org/rehabilitation-measures/6-minute-walk-test.
- [Background] Bohannon RW, Bubela DJ, Wang YC, Magasi SS, Gershon RC. Six-Minute Walk Test Vs. Three-Minute Step Test for Measuring Functional Endurance. J Strength Cond Res. 2015 Nov;29(11):3240-4. doi: 10.1519/JSC.0000000000000253. PMID 24077375